CLINICAL TRIAL: NCT01085045
Title: A Randomized, Double-Blind (Test Products and Placebo), Chronic Dosing (7 Days), Four-Period, Eight-Treatment, Placebo-Controlled, Incomplete Block, Cross-Over, Multi-Center Study to Assess Efficacy and Safety of Two Doses of PT003, Two Doses of PT005 and One Dose of PT001 in Patients With Moderate to Very Severe COPD, Compared With Foradil® Aerolizer® (12 μg, Open-Label) and Spiriva® Handihaler® (18 μg, Open-Label) as Active Controls
Brief Title: Study to Evaluate the Efficacy, Safety and Pharmacokinetics of PT001, PT003, and PT005 Following Chronic Dosing (7 Days) in Patients With Moderate to Very Severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PT0031002
Record Dates: First submitted 2010-03-09; First posted 2010-03-11 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Inhaled PT003 (Dose 1) (Experimental): PT003 MDI Dose 1
  Interventions: Drug: PT003 MDI
- Inhaled PT003 (Dose 2) (Experimental): PT003 MDI Dose 2
  Interventions: Drug: PT003 MDI
- Inhaled PT005 (Dose 1) (Experimental): PT005 MDI Dose 1
  Interventions: Drug: PT005 MDI
- Inhaled PT005 (Dose 2) (Experimental): PT005 MDI Dose 2
  Interventions: Drug: PT005 MDI
- Inhaled Placebo (Placebo Comparator): Placebo MDI
  Interventions: Drug: Placebo MDI
- Tiotropium bromide 18 μg (Spiriva Handihaler®) (Active Comparator): Tiotropium Bromide inhalation powder
  Interventions: Drug: Tiotropium bromide 18 μg (Spiriva Handihaler®)
- Formoterol Fumarate 12 μg (Foradil® Aerolizer®) (Active Comparator): Formoterol fumarate inhalation powder 12 μg
  Interventions: Drug: Formoterol Fumarate 12 μg (Foradil® Aerolizer®)
- Inhaled PT001 (Dose 1) (Experimental): PT001 MDI Dose 1
  Interventions: Drug: PT001 MDI

INTERVENTIONS:
Drug: PT003 MDI — Inhaled PT003 MDI administered as two puffs BID for 7 days
  Arms: Inhaled PT003 (Dose 1); Inhaled PT003 (Dose 2)
Drug: PT005 MDI — Inhaled PT005 MDI administered as two puffs BID for 7 days
  Arms: Inhaled PT005 (Dose 1); Inhaled PT005 (Dose 2)
Drug: Placebo MDI — Inhaled placebo administered as two puffs BID for 7 days
  Arms: Inhaled Placebo
Drug: Tiotropium bromide 18 μg (Spiriva Handihaler®) — Inhaled tiotropium bromide 18 μg (Spiriva Handihaler®) administered QD for 7 days
  Arms: Tiotropium bromide 18 μg (Spiriva Handihaler®)
Drug: Formoterol Fumarate 12 μg (Foradil® Aerolizer®) — Inhaled formoterol fumarate 12 μg (Foradil® Aerolizer®) administered BID for 7 days
  Arms: Formoterol Fumarate 12 μg (Foradil® Aerolizer®)
Drug: PT001 MDI — Inhaled PT001 MDI administered as two puffs BID for 7 days
  Arms: Inhaled PT001 (Dose 1)

SUMMARY:
The purpose of this study is to evaluate, after 1 week of dosing, the efficacy and safety of PT003 compared with its individual components (PT001 and PT005), placebo and two active comparators to demonstrate superiority of the combination to its components, and to assess the relative contribution of the components compared with placebo, in patients with moderate to very severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* 40 - 80 years of age
* Clinical history of COPD with airflow limitation that is not fully reversible
* Females of non-child bearing potential or females of child bearing potential with negative pregnancy test; and acceptable contraceptive methods
* Current/former smokers with at least a 10 pack-year history of cigarette smoking
* A measured post- bronchodilator FEV1/FVC ratio of < or = 0.70
* A measured post- bronchodilator FEV1 > or = 750ml or 30% predicted and < or = 80% of predicted normal values
* Able to change COPD treatment as required by protocol

Exclusion Criteria:

* Women who are pregnant or lactating
* Primary diagnosis of asthma
* Alpha-1 antitrypsin deficiency as the cause of COPD
* Active pulmonary diseases
* Prior lung volume reduction surgery
* Abnormal chest X-ray (or CT scan) not due to the presence of COPD
* Hospitalized due to poorly controlled COPD within 3 months of Screening
* Clinically significant medical conditions that preclude participation in the study (e.g. clinically significant abnormal ECG, uncontrolled hypertension, glaucoma, symptomatic prostatic hypertrophy)
* Cancer that has not been in complete remission for at least 5 years
* Treatment with investigational study drug or participation in another clinical trial or study within the last 30 days or 5 half lives

Other protocol defined inclusion/exclusion criteria may apply

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, M.D., Study Director — Pearl Therapeutics, Inc.
Locations (16):
- United States (4):
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - American Health Research, Charlotte, North Carolina
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Spartanburg Medical Research, Spartanburg, South Carolina
- Australia (8):
  - Austrials, Caringbah, New South Wales
  - Woolcock, Glebe, New South Wales
  - Austrials, Hornsby, New South Wales
  - Austrials, Auchenflower, Queensland
  - Q-Pharm, Herston, Queensland
  - Respiratory Research Foundation - Burnside War Memorial Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Lung Institute of WA, Nedlands, Western Australia
- New Zealand (4):
  - Greenlane Clinical Centre, Epsom, Auckland
  - NZ Respiratory & Sleep Institute, Greenlane East, Auckland
  - Waikato Hospital, Hamilton, Waikato Region
  - P3 Research, Crofton Downs, Wellington Region

REFERENCES:
- [Derived] Reisner C, Fabbri LM, Kerwin EM, Fogarty C, Spangenthal S, Rabe KF, Ferguson GT, Martinez FJ, Donohue JF, Darken P, St Rose E, Orevillo C, Strom S, Fischer T, Golden M, Dwivedi S. A randomized, seven-day study to assess the efficacy and safety of a glycopyrrolate/formoterol fumarate fixed-dose combination metered dose inhaler using novel Co-Suspension Delivery Technology in patients with moderate-to-very severe chronic obstructive pulmonary disease. Respir Res. 2017 Jan 6;18(1):8. doi: 10.1186/s12931-016-0491-8. PMID 28061907

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at 16 sites in Australia, New Zealand and the US from 24 March 2010 -28 October 2010. The entire study period was a maximum of 20 weeks. Chronic dosing (7 days), 4-period, 8-treatment, incomplete block, cross-over conducted in two parts.
Pre-assignment Details: Part A: 4-period, 8-treatment, incomplete block cross-over. Subjects randomized to 1 of 48 sequences, each subject received 4 of 8 possible treatments. Part B: 4-period, 4-treatment, full cross-over. Each subject randomized to 1 of 24 sequences and each sequence was assigned to at least 1 subject.
Groups:
- Overall Study: Sentinel patients were the first 4 patients enrolled to receive one week of treatment with either GFF MDI 72/9.6mcg, GFF MDI 36/9.6 mcg, GP MDI 36 mcg or FF MDI 9.6 mcg because this was the first time GFF MDI was administered to patients with COPD, the sentinel patients provided additional assurance of safety.9.6
Period: Part A
Arm/Group | Overall Study
Started | 122
GFF MDI 72/9.6mcg | 40
GFF MDI 36/9.6 µg (PT003) | 42
GP MDI 36 µg (PT001) | 40
Spiriva 18 µg | 58
FF MDI 9.6 µg (PT005) | 20
FF MDI 7.2 µg (PT005) | 21
Placebo MDI | 5
Foradil 12 µg | 14
Completed | 104
Not Completed | 18
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 6
Not completed — Protocol Violation | 1
Not completed — Protocol Specified Criteria | 7
Period: Part B
Arm/Group | Overall Study
Started | 104
GFF MDI 72/9.6mcg (PT003) | 0
GFF MDI 36/9.6 µg | 0
Spiriva 18 µg | 0
FF MDI 9.6 µg (PT005) | 43
FF MDI 7.2 µg (PT005) | 43
Placebo MDI | 47
Foradil 12 µg | 41
GP MDI 36 µg (PT001) | 0
Completed | 89
Not Completed | 15
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Specified Criteria | 6
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 6

BASELINE CHARACTERISTICS:
Population: Analysis Population included all randomized participants. 118 plus 4 sentinel patients to make 122.
Groups:
- All Subjects: All Baseline Subjects
Arm/Group | All Subjects
Number analyzed (Participants) | 122
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.4 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 69

OUTCOME MEASURES:

1. Primary Outcome: FEV1 AUC 0-12 on Day 7
Description: Forced Expiratory Volume in One Second (FEV1) Area Under the Curve (AUC) 0-12 (normalized) relative to baseline FEV1 following 7-day dose administration
Time Frame: "Pre-dose, 15 minutes, 30 minutes, 1, 2, 4, 6, 8, 10, 11.5, and 12 hours post-dose on Day 7
Population: Modified Intent to Treat (MITT) Population - not including the 4 sentinel patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- GFF MDI 72/9.6 μg: GFF MDI 72/9.6 μg (PT003)
- GFF MDI 36/9.6 μg: GFF MDI 36/9.6 μg (PT003)
- GP MDI 36 μg: GP MDI 36 μg (PT001)
- Spiriva 18 μg: Spiriva 18 μg
- FF MDI 9.6 μg: FF MDI 9.6 μg (PT005)
- FF MDI 7.2 μg: FF MDI 7.2 μg (PT005)
- Foradil 12 μg: Foradil 12 μg
Arm/Group | GFF MDI 72/9.6 μg | GFF MDI 36/9.6 μg | GP MDI 36 μg | Spiriva 18 μg | FF MDI 9.6 μg | FF MDI 7.2 μg | Foradil 12 μg
Number analyzed (Participants) | 37 | 38 | 35 | 53 | 55 | 58 | 53
Liters | 1.537 [1.499 to 1.575] | 1.529 [1.492 to 1.567] | 1.429 [1.389 to 1.469] | 1.434 [1.401 to 1.467] | 1.421 [1.386 to 1.455] | 1.413 [1.379 to 1.446] | 1.437 [1.401 to 1.472]

2. Secondary Outcome: Peak Change From BL in FEV1 on Day 1
Description: Peak change from Baseline in FEV1 on Day 1
Time Frame: Day 1
Population: MITT Population - not including the 4 sentinel patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI 72/9.6 μg | GFF MDI 36/9.6 μg | GP MDI 36 μg | Spiriva 18 μg | FF MDI 9.6 μg | FF MDI 7.2 μg | Foradil 12 μg
Number analyzed (Participants) | 38 | 39 | 38 | 56 | 58 | 63 | 54
Liters | 0.370 [0.325 to 0.416] | 0.357 [0.312 to 0.401] | 0.289 [0.243 to 0.335] | 0.266 [0.229 to 0.304] | 0.308 [0.269 to 0.348] | 0.310 [0.273 to 0.348] | 0.299 [0.258 to 0.340]

3. Secondary Outcome: Peak Change From BL in FEV1 on Day 7
Description: Peak change from Baseline (BL) in FEV1 on Day 7
Time Frame: Day 7
Population: MITT Population - not including the 4 sentinel patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI 72/9.6 μg | GFF MDI 36/9.6 μg | GP MDI 36 μg | Spiriva 18 μg | FF MDI 9.6 μg | FF MDI 7.2 μg | Foradil 12 μg
Number analyzed (Participants) | 38 | 39 | 38 | 53 | 58 | 61 | 54
Liters | 0.438 [0.396 to 0.481] | 0.440 [0.398 to 0.481] | 0.313 [0.270 to 0.356] | 0.298 [0.262 to 0.335] | 0.337 [0.300 to 0.374] | 0.330 [0.294 to 0.366] | 0.356 [0.317 to 0.395]

4. Secondary Outcome: Peak Change From BL in Inspiratory Capacity on Day 1
Description: Peak change from Baseline in Inspiratory Capacity (IC) on Day 1
Time Frame: Day 1
Population: MITT Population - not including the 4 sentinel patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI 72/9.6 μg | GFF MDI 36/9.6 μg | GP MDI 36 μg | Spiriva 18 μg | FF MDI 9.6 μg | FF MDI 7.2 μg | Foradil 12 μg
Number analyzed (Participants) | 38 | 39 | 38 | 56 | 58 | 63 | 54
Liters | 0.495 [0.411 to 0.579] | 0.411 [0.330 to 0.493] | 0.430 [0.346 to 0.514] | 0.347 [0.278 to 0.416] | 0.362 [0.290 to 0.433] | 0.352 [0.283 to 0.420] | 0.374 [0.299 to 0.449]

5. Secondary Outcome: Peak Change From BL IC on Day 7
Description: Peak Change from Baseline Inspiratory Capacity on following 7-day dose administration
Time Frame: Day 7
Population: MITT Population - not including the 4 sentinel patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI 72/9.6 μg | GFF MDI 36/9.6 μg | GP MDI 36 μg | Spiriva 18 μg | FF MDI 9.6 μg | FF MDI 7.2 μg | Foradil 12 μg
Number analyzed (Participants) | 37 | 39 | 38 | 53 | 58 | 61 | 54
Liters | 0.409 [0.327 to 0.491] | 0.438 [0.359 to 0.516] | 0.331 [0.249 to 0.412] | 0.314 [0.244 to 0.383] | 0.359 [0.289 to 0.430] | 0.376 [0.307 to 0.444] | 0.393 [0.319 to 0.466]

6. Secondary Outcome: Time to Onset of Action >=10% Improvement in FEV1 on Day 1
Description: Time to Onset of Action where the improvement in FEV1 on Day 1 was >=10%
Time Frame: Day 1
Population: MITT Population - not including the 4 sentinel patients.
Measure: Number; unit: Participants
Arm/Group | GFF MDI 72/9.6 μg | GFF MDI 36/9.6 μg | GP MDI 36 μg | Spiriva 18 μg | FF MDI 9.6 μg | FF MDI 7.2 μg | Foradil 12 μg
Number analyzed (Participants) | 36 | 39 | 37 | 54 | 57 | 61 | 50
Participants
  15 Minutes | 22 | 20 | 14 | 22 | 37 | 34 | 30
  30 Minutes | 5 | 7 | 10 | 4 | 10 | 12 | 6
  60 Minutes | 4 | 6 | 3 | 7 | 4 | 4 | 6
  120 Minutes | 2 | 1 | 4 | 5 | 0 | 2 | 3
  No onset | 3 | 5 | 6 | 16 | 6 | 9 | 5

7. Secondary Outcome: Percentage of Patients Achieving >=12% Improvement in FEV1 on Day 1
Description: Time to Onset of Action where the improvement in FEV1 on Day 1 was >= 12%
Time Frame: Day 1
Population: MITT Population - not including the 4 sentinel patients.
Measure: Number; unit: Percentage of Participants
Arm/Group | GFF MDI 72/9.6 μg | GFF MDI 36/9.6 μg | GP MDI 36 μg | Spiriva 18 μg | FF MDI 9.6 μg | FF MDI 7.2 μg | Foradil 12 μg
Number analyzed (Participants) | 38 | 39 | 38 | 56 | 58 | 63 | 54
Percentage of Participants | 86.84 | 87.18 | 73.68 | 66.07 | 84.48 | 82.54 | 85.19

8. Secondary Outcome: Change in Morning Pre-dose FEV1 on Day 7
Description: Change from Baseline in morning pre-dose FEV1 on Day 7
Time Frame: Day 7
Population: MITT Population - not including the 4 sentinel patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI 72/9.6 μg | GFF MDI 36/9.6 μg | GP MDI 36 μg | Spiriva 18 μg | FF MDI 9.6 μg | FF MDI 7.2 μg | Foradil 12 μg
Number analyzed (Participants) | 38 | 39 | 38 | 53 | 58 | 61 | 54
Liters | 0.193 [0.148 to 0.237] | 0.170 [0.126 to 0.213] | 0.097 [0.052 to 0.142] | 0.097 [0.058 to 0.136] | 0.064 [0.024 to 0.103] | 0.073 [0.034 to 0.111] | 0.101 [0.060 to 0.142]

9. Secondary Outcome: 12 hr Post-dose Trough FEV1 on Day 7
Description: 12 hour post-dose trough Forced Expiratory Volume in 1 second on Day 7
Time Frame: Day 7
Population: MITT Population - not including the 4 sentinel patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MDI 72/9.6 μg | GFF MDI 36/9.6 μg | GP MDI 36 μg | Spiriva 18 μg | FF MDI 9.6 μg | FF MDI 7.2 μg | Foradil 12 μg
Number analyzed (Participants) | 37 | 38 | 35 | 53 | 55 | 58 | 53
Liters | 1.405 [1.358 to 1.453] | 1.441 [1.395 to 1.488] | 1.383 [1.333 to 1.432] | 1.398 [1.357 to 1.439] | 1.349 [1.306 to 1.393] | 1.378 [1.336 to 1.419] | 1.358 [1.314 to 1.402]

10. Secondary Outcome: Change From BL in Mean Morning Pre-dose Daily Peak Flow Rate on Day 7
Description: Change from BaseLine in mean morning pre-dose daily peak flow rate on Day 7
Time Frame: Day 7
Population: MITT Population - not including the 4 sentinel patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters / Minute
Arm/Group | GFF MDI 72/9.6 μg | GFF MDI 36/9.6 μg | GP MDI 36 μg | Spiriva 18 μg | FF MDI 9.6 μg | FF MDI 7.2 μg | Foradil 12 μg
Number analyzed (Participants) | 38 | 39 | 38 | 54 | 56 | 60 | 52
Liters / Minute | 30.263 [21.479 to 39.046] | 28.152 [19.756 to 36.547] | 16.439 [7.620 to 25.259] | 11.817 [4.316 to 19.317] | 12.424 [4.593 to 20.256] | 10.211 [2.692 to 17.730] | 13.426 [5.426 to 21.426]

11. Secondary Outcome: Change From BL in Mean Morning Post-dose Daily Peak Flow Rate on Day 7
Description: Change from BaseLine in mean morning post-dose daily peak flow rate on Day 7
Time Frame: Day 7
Population: MITT Population - not including the 4 sentinel patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters / Minute
Arm/Group | GFF MDI 72/9.6 μg | GFF MDI 36/9.6 μg | GP MDI 36 μg | Spiriva 18 μg | FF MDI 9.6 μg | FF MDI 7.2 μg | Foradil 12 μg
Number analyzed (Participants) | 38 | 39 | 38 | 54 | 56 | 60 | 52
Liters / Minute | 56.666 [47.631 to 65.700] | 53.411 [44.600 to 62.221] | 33.652 [24.553 to 42.750] | 27.668 [19.742 to 35.594] | 41.287 [33.105 to 49.468] | 38.712 [30.799 to 46.624] | 39.132 [30.761 to 47.502]

12. Secondary Outcome: Change From BL in Mean Evening Pre-dose Daily Peak Flow Rate on Day 7
Description: Change from BaseLine in mean evening pre-dose daily peak flow rate on Day 7
Time Frame: Day 7
Population: MITT Population - not including the 4 sentinel patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters / Minute
Arm/Group | GFF MDI 72/9.6 μg | GFF MDI 36/9.6 μg | GP MDI 36 μg | FF MDI 9.6 μg | FF MDI 7.2 μg | Foradil 12 μg
Number analyzed (Participants) | 38 | 39 | 38 | 56 | 60 | 52
Liters / Minute | 35.0945 [25.888 to 44.302] | 30.817 [21.713 to 39.920] | 18.487 [9.034 to 27.939] | 17.190 [9.029 to 25.350] | 14.805 [6.800 to 22.810] | 17.789 [9.383 to 26.194]

13. Secondary Outcome: Change From BL in Mean Evening Post-dose Daily Peak Flow Rate on Day 7
Description: Change from BaseLine in mean evening post-dose daily peak flow rate on Day 7
Time Frame: Day 7
Population: MITT Population - not including the 4 sentinel patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters / Minute
Arm/Group | GFF MDI 72/9.6 μg | GFF MDI 36/9.6 μg | GP MDI 36 μg | Spiriva 18 μg | FF MDI 9.6 μg | FF MDI 7.2 μg | Foradil 12 μg
Number analyzed (Participants) | 38 | 39 | 38 | 51 | 56 | 59 | 52
Liters / Minute | 53.863 [43.924 to 63.802] | 58.326 [48.553 to 68.099] | 36.637 [26.685 to 46.589] | 24.253 [15.172 to 33.335] | 41.395 [32.252 to 50.538] | 37.192 [28.251 to 46.132] | 39.323 [30.024 to 48.621]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed consent through Visit 10/Final Visit (7-14 days post final dose).
Description: Serious Adverse Events (SAE) were captured from the time subjects sign the ICF through the final visit or premature discontinuation visit up to 30 days following the last dose of study drug. Safety population included all participants who were randomized to treatment and received at least one dose of one study treatment.
Groups:
- GP/FF MDI 72/9.6 μg: GP/FF MDI 72/9.6 μg (PT003)
- GP/FF MDI 36/9.6 μg: GP/FF MDI 36/9.6 μg (PT003)
- Spiriva: Handihaler 18 μg
- Placebo: Placebo MDI
- Foradil Aerolizer: Foradil Aerolizer 12 μg
Arm/Group | GP/FF MDI 72/9.6 μg | GP/FF MDI 36/9.6 μg | GP MDI 36 μg | Spiriva | FF MDI 9.6 μg | FF MDI 7.2 μg | Placebo | Foradil Aerolizer
Serious Adverse Events (participants affected / at risk) | 0/41 | 1/43 | 0/41 | 2/58 | 1/64 | 2/64 | 0/52 | 0/55
Other Adverse Events (participants affected / at risk) | 14/41 | 17/43 | 10/41 | 9/58 | 5/64 | 4/64 | 4/52 | 7/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP/FF MDI 72/9.6 μg (N=41) | GP/FF MDI 36/9.6 μg (N=43) | GP MDI 36 μg (N=41) | Spiriva (N=58) | FF MDI 9.6 μg (N=64) | FF MDI 7.2 μg (N=64) | Placebo (N=52) | Foradil Aerolizer (N=55)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foreign Body Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP/FF MDI 72/9.6 μg (N=41) | GP/FF MDI 36/9.6 μg (N=43) | GP MDI 36 μg (N=41) | Spiriva (N=58) | FF MDI 9.6 μg (N=64) | FF MDI 7.2 μg (N=64) | Placebo (N=52) | Foradil Aerolizer (N=55)
Dry Mouth (Gastrointestinal disorders) | 8 (10) | 3 (5) | 6 (7) | 5 (6) | 3 (4) | 3 (4) | 1 (1) | 3 (4)
Headache (Nervous system disorders) | 5 (6) | 5 (19) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Tremor (Nervous system disorders) | 1 (1) | 6 (8) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent its opinions, or the opinions of the publication committee, if these differ with the proposed publication.